CLINICAL TRIAL: NCT06636786
Title: Prevention/Reduction of ASRs and PTSD to Sustain Civilian Performance With Sublingual Cyclobenzaprine HCl (TNX-102 SL) - (Optimizing Acute Stress Reaction Interventions With TNX-102 SL - OASIS)
Brief Title: Prevention/Reduction of ASRs and PTSD to Sustain Civilian Performance With Sublingual Cyclobenzaprine HCl (TNX-102 SL)
Acronym: OASIS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Tonix Pharmaceuticals, Inc. (Industry); Mclean Hospital (Other); Cooper University Health Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 23-0711
Record Dates: First submitted 2024-09-05; First posted 2024-10-15 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Acute Stress Reaction; Acute Stress Disorder; Neurocognitive Function; Post-traumatic Stress
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute | interventions — cyclobenzaprine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cyclobenzaprine HCl (Experimental): Participants will be instructed to take a half dose (equivalent to 1 tablet, 2.8 mg) of Cyclobenzaprine HCl in the ED as part of enrollment procedures. If the time between the first half dose and the planned bedtime of the participant is less than 6 hours, participants will be instructed to take 1 tablet (half dose) the first night at bedtime. If the time between the first half dose and planned bedtime of the participant is greater than or equal to 6 hours, then participants will be instructed to take a full dose (equivalent to 2 tablets) the first night. Over the following 13 days, all participants will be instructed to take a full dose of the study drug at bedtime. Each participant will receive 29 tablets and take either 28 or 29 tablets total for the duration of study participation.
  Interventions: Drug: Cyclobenzaprine HCl
- Placebo (Placebo Comparator): Participants will be instructed to take a half dose (equivalent to 1 tablet, 2.8 mg) of placebo in the ED as part of enrollment procedures. The placebo is the same formulation as active except the Cyclobenzaprine HCl content is replaced by Mannitol to maintain the same tablet weight and dimensions. If the time between the first half dose and the planned bedtime of the participant is less than 6 hours, participants will be instructed to take 1 tablet (half dose) the first night at bedtime. If the time between the first half dose and planned bedtime of the participant is greater than or equal to 6 hours, then participants will be instructed to take a full dose (equivalent to 2 tablets) the first night. Over the following 13 days, all participants will be instructed to take a full dose of the study drug at bedtime. Each participant will receive 29 tablets and take either 28 or 29 tablets total for the duration of study participation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyclobenzaprine HCl — TNX-102 SL (cyclobenzaprine HCl sublingual tablets) taken sublingually (under the tongue) in the ED and each day at bedtime for a total of 2 weeks.
  Other Names: TNX-102 SL
  Arms: Cyclobenzaprine HCl
Drug: Placebo — Placebo sublingual tablets taken sublingually (under the tongue) in the ED and each day at bedtime for a total of 2 weeks.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This study will examine the safety and efficacy of TNX-102 SL to reduce ASR symptoms and behavioral changes among patients presenting to the emergency department (ED) after motor vehicle collision (MVC). Specifically, the investigators will perform the Optimizing Acute Stress reaction Interventions with TNX-102 SL (OASIS) Trial, a double-blind placebo-controlled randomized clinical trial (RCT) to determine if TNX-102 SL initiated in the ED in the hours after MVC to high risk individuals, treats/reduces acute stress reaction (ASR)/acute stress disorder (ASD) symptoms (primary outcome), improves neurocognitive function, and prevents/reduces posttraumatic stress (PTS) symptoms (secondary outcomes) long term. 180 participants will be randomized, receive study drug in ED and be discharged with a 2-week drug supply. Prior to initial dose of study drug administration, and during the hours, days, and weeks after participants will receive serial longitudinal assessments of psychological and somatic symptoms, neurocognitive function, and adverse events.

DETAILED DESCRIPTION:
U.S. military personnel are exposed to life-threatening traumatic events (e.g., intense firefights with multiple casualties) that result in acute stress reaction (ASR) symptoms (ICD-10) and posttraumatic stress (PTS). Similarly, acute and persistent stress symptoms, and related adverse posttraumatic neuropsychiatric sequelae, are also very common and cause a tremendous burden of suffering in civilian populations following exposure to life-threatening traumatic events (e.g., motor vehicle collision, violent or accidental death of a loved one, and assault). TNX-102 SL (cyclobenzaprine HCl sublingual tablet) is being developed for the management of fibromyalgia (FM), and post-traumatic stress disorder (PTSD) by Tonix Pharmaceuticals, Inc; the FM program is in mid-Phase 3 development and PTSD is Phase 3 ready. In previous PTSD and fibromyalgia studies, TNX-102 SL has demonstrated the ability to improve sleep quality, which, based on published clinical studies of fear memory and stress responsiveness, has been shown to play a significant role in stress recovery. To date, TNX-102 SL has undergone an intense nonclinical and clinical development including Phase 1, 2, and 3 studies that assessed safety in over 1,180 subjects. TNX-102 SL is an extremely promising agent to reduce ASR symptoms and related behavioral changes, to enhance resilience and improve warfighter performance, and to reduce the frequency and severity of persistent/chronic PTS symptoms. The results of this study will ultimately provide military personnel, veterans, and civilians with an important new treatment option that, when administered in the early aftermath of traumatic stress exposure, can improve recovery, job performance, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years and ≤ 55 years of age
* Admitted to ED within 24 hours of MVC
* Anticipated to be discharged home from the ED
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Consent to receive unencrypted communications
* Has a smartphone with continuous service for ≥ 1 year
* Has a personal email address they regularly access
* Able to speak and read English
* PTS prediction tool risk score ≥ 16 in the ED
* Pain severity in the ED ≥ 4 (0-10 numeric rating scale)
* People who are not of childbearing potential (e.g., hysterectomy, bilateral oophorectomy, or confirmed postmenopausal for at least last 12 consecutive months)
* People with the capacity to conceive a pregnancy must agree to employ a highly effective form of birth control throughout the first 21 days of study participation (e.g., oral, injected, transdermal, or implanted hormonal methods of contraception for at least one full menstrual cycle prior to study drug administration; placement of an intrauterine device (IUD) or intrauterine system (IUS); or double barrier methods such as condoms and diaphrams)

Exclusion Criteria:

* Substantial comorbid injury (e.g., long bone fracture)
* People of childbearing potential who are pregnant, breastfeeding, planning to become pregnant, or not using a highly effective form of contraception (e.g., implants, intrauterine devices (IUDs), tubal ligation, hormonal birth control pills, patches, vaginal rings, or injections) during their participation
* Prisoner status
* Any chronic daily opioid use prior to MVC
* Active psychosis, suicidal ideation, or homicidal ideation
* Plans for hospital admission
* History of arrhythmias, heart block or conduction disturbances, congestive heart failure
* Currently in the acute recovery phase of myocardial infarction
* Hypersensitivity to cyclobenzaprine or the excipient in TNX-102 SL or placebo formulations
* History of urinary retention, angle-closure glaucoma, increased intraocular pressure, or hyperthyroidism (TSH < lower limit of normal)
* Concomitant use of monoamine oxidase (MAO) inhibitors or within 14 days after their discontinuation due to risk of potential fatal drug-drug interactions
* Current or planned use of the following prohibited concomitant medications during study participation: anticholinergic medications, guanethidine, selective serotonin reuptake inhibitors (SSRIs) , serotonin norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants (TCAs), tramadol, bupropion, meperidine, verapamil, MAO inhibitors, anticholinergic medications, guanethidine, potent cytochrome P450 subtype 3A4 inhibitor, St. John's wort, or other prohibited concomitant medications listed in section 5.6 of protocol
* Any hepatic impairment or renal disease (defined as aspartate transaminase (AST) or alanine transaminase (ALT) > 3 times the upper limit of normal) or renal disease (defined as glomerular filtration rate (GFR) ≤ 80 mL/min)
* Lacking capacity to provide informed consent (receipt of sedative, hypnotic agent making the patient non-decisional for consent)
* Any other history or condition that would, in the site investigator's judgement, indicate that the patient would very likely be non-compliant with the study or unsuitable for the study (e.g., might interfere with the study, confound interpretation, or endanger patient)
* Elevated baseline blood pressure defined as systolic blood pressure ≥ 170 mmHg or diastolic blood pressure ≥ 100 mmHg and or elevated heart rate of ≥115
* Abnormal baseline ECG as defined as: QRS duration ≥ 120 ms; QTc > 460 ms; not in sinus rhythm; or 1st, 2nd, or 3rd degree heart block indicated
* Substance or alcohol use disorder, bipolar disorder, or schizophrenia
* History of severe or unexplained oral, or oropharyngeal swelling or edema

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in ASD Score | Week 1, 3 after MVC
  Individuals are asked to complete the 14-item Acute Stress Disorder Scale (ASDS) self-report inventory where each item is rated on a 5-point scale (0= Not at all; 1= Mildly; 2= Medium; 3= Quite a bit; 4= Very Much) that indexes acute stress disorder (ASD). Range of possible total scores is 0-56, with higher total scores indicating greater acute stress symptoms.

SECONDARY OUTCOMES:
Median reaction time of correct responses (general cognitive function) | Min 30, Hour 1, 6, 12, Day 1, 2, 3, Week 1, 2, 3, 5, 6, 8, 11, 12 after MVC
  General cognitive function will be assessed using the Test My Brain Digit Symbol Matching Test. Participants will be asked to match symbols and numbers using a symbol-number key shown on screen. General cognitive function is assessed via measuring median reaction time of correct responses (medianRTc) to 'test' trials. Range for medianRTc (ms) is 0-30000.
Median reaction time of correct responses (procedural reaction time) | Min 30, Hour 1, 6, 12, Day 1, 2, 3, Week 1, 2, 3, 5, 6, 8, 11, 12 after MVC
  Procedural reaction time will be assessed using the Test My Brain Choice Reaction Time Test. Participants see a set of three arrows, where one arrow is a different color from the rest. The participant presses left or right to indicate the direction of the odd colored arrow. Reaction time is assessed via measuring median reaction time of correct responses (medianRTc) to 'test' trials. Range for medianRTc (ms) is 0-5000.
Proportion of targets correctly identified (visuospatial processing and attention) | Min 30, Hour 1, 6, 12, Day 1, 2, 3, Week 1, 2, 3, 5, 6, 8, 11, 12 after MVC
  Visuospatial processing and attention will be assessed using the Test My Brain Multiple Object Tracking Test. In this test of visuospatial processing and attention, participants have to track a set of target circles around the screen (amidst a field of distractors) that move at increasing speed with each trial. Once the circles stop moving, participants select which were targets must identify targets instead of distractors. Visuospatial processing and attention are assessed via the proportion of targets correctly identified. Range for measure is 0-1.
d-prime identification (psychomotor vigilance) | Min 30, Hour 1, 6, 12, Day 1, 2, 3, Week 1, 2, 3, 5, 6, 8, 11, 12 after MVC
  Psychomotor vigilance will be assessed via the Test My Brain Gradual Onset Continuous Performance Test. In this task, participants monitor a stream of city and mountain images that rapidly fade from one to the next with no interstimulus interval. Participants are asked to press/touch for each city image and to withhold for each mountain image. Vigilance is assessed via measuring d-prime for identification of each city image, a signal detection-based measure that takes into account both hits and false alarms to provide an unbiased estimate of performance where higher values reflect better performance. Response inhibition is defined as the suppression of actions that are inappropriate in a given context. Response inhibition is assessed using results from the above, by measuring the number of commission errors (failure to withhold responses) where most positive scores reflect more impulsive responding. Range for measure is -4.2279 - 4.2279.
Change in Pain Symptom Score | Baseline, Week 1, 3, 6, 12 after MVC
  The Regional Pain Scale (RPS) will be used to assess the extent of body pain. 13 items will be scored on a 0-10 pain scale where 0 is no pain and 10 is severe pain. Range of possible total scores is 0-130, with higher total scores indicative of greater pain symptoms
Change in Depressive Symptoms Score | Baseline, Week 1, 3, 6, 12 after MVC
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form 8b; an 8-item scale, and one question from the PROMIS Depression Item Bank will be aggregated/combined to assess depression. Each item is scored on a 5-point scale where 0 is "none of the time" and 5 means "all or almost all of the time". Range of possible total scores is 0-45, with higher total scores indicative of greater depressive symptoms.
Change in Somatic Symptom Score | Baseline, Week 1, 3, 6, 12 after MVC
  The Pennebaker Inventory of Limbic Languidness (PILL) assesses the frequency of common physical symptoms and sensations. We will use a version with adapted response options for greater consistency across measures, greater precision in response levels, and to allow administration via self-report. 20 items will be scored on a 0-10 scale where 0 is "no problem" and 10 means "major problem". Range of possible total scores is 0-200, with higher total scores indicative of greater somatic symptoms.
Change in PTSD Symptoms | Baseline, Week 1, 3, 6, 12 after MVC
  The PTSD Checklist for DSM-5 (PCL-5) assesses PTSD symptoms as defined by the Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5). 20 items will be scored on a five-point scale ranging from 0 ("not at all") to 4 ("extremely"). Range of possible total scores is 0-80, with higher total scores indicative of greater PTSD symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel McLean, MD, Principal Investigator — University of North Carollina at Chapel Hill; Christopher Jones, MD, Principal Investigator — Cooper University Health Care
Locations (6):
- United States (6):
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Massachusetts Chan Medical School (Umass Memorial Medical Center), Worcester, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 12 months following publication and continuing for 36 months.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.